CLINICAL TRIAL: NCT03996278
Title: Comparison Thymoglobulin® Versus Grafalon® in Renal Transplantation - Spiesser Group (Retro/Prospective Study) I
Brief Title: Comparison Thymoglobulin® and Grafalon®
Acronym: THYGRET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0018
Record Dates: First submitted 2019-05-28; First posted 2019-06-24 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Renal Transplantation
Keywords: THYMOGLOBULINE®; GRAFALON®
MeSH Terms: interventions — thymoglobulin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients in the Grafalon group: Patients in the Grafalon group (n=150) will be followed prospectively and data prospectively collected thanks to the Astre database
  Interventions: Other: Grafalon
- Patients in the Thymoglobulin group: Patients in the thymoglobulin group (n=150) will be selected and analyzed retrospectively from the Astre database
  Interventions: Other: Grafalon

INTERVENTIONS:
Other: Grafalon — None interventional study but there are two groups
  Other Names: Thymoglobulin

SUMMARY:
This is a prospective, multicenter, observational, non -interventional study with comparison with an historical cohort Investigators will compare the efficacy and safety of Thymoglobulin (Sanofi-Aventis) versus Grafalon (Neovii, previously ATG-Fresenius) in renal transplantation by evaluating patient survival, graft survival, delayed graft function, acute rejection, DSA occurrence and toxicities, various infections including CMV and BK virus incidence, MACE (major cardiac adverse event) and cancer.

Investigators will also compare cumulative treatment and follow up costs and other key criteria available in the ASTRE database.

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational, non -interventional study with comparison with an historical cohort Investigators will compare the efficacy and safety of Thymoglobulin (Sanofi-Aventis) versus Grafalon (Neovii, previously ATG-Fresenius) in renal transplantation by evaluating patient survival, graft survival, delayed graft function, acute rejection, DSA occurrence and toxicities, various infections including CMV and BK virus incidence, MACE (major cardiac adverse event) and cancer.

Investigators will also compare cumulative treatment and follow up costs and other key criteria available in the ASTRE database.

Justification for a non-interventional study: in the study the medicinal products will be prescribed in the usual manner in accordance with the terms of the marketing authorisation. The assignment of the patient to the product is not decided in advance by a trial protocol but falls within current practice of the centre and the prescription of the medicine is clearly separated from the decision to include the patient in the study. No additional diagnostic or monitoring procedures are applied to the patients and epidemiological methods are used for the analysis of collected data.

ELIGIBILITY:
Inclusion Criteria:

* For the Grafalon prospective group: all first 11-12 patients from the 13 transplant centres receiving Grafalon according to the local practice
* For the Thymoglobulin group: a group of 130 patients matched for:

age (donor and recipient) gender indication (immunological indication versus DFG) CMV status

Exclusion Criteria:

* Patient younger than 18 years old
* Living donor
* Donor after cardiac death (because the Maastricht 3 donors are authorized recently in France)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received or are receiving induction ATGs at the time of transplantation and whose data are collected from the ASTRE base in the 13 renal transplant centrers participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-05-22 (Estimated); Study Completion 2021-11-22 (Estimated)

PRIMARY OUTCOMES:
Comparison adverse events of the 2 ATGs and data collected thanks to the ASTRE database | During one year
  All events: Death, graft loss, acute rejection, DGF, de novo DSA Severe infection (SAE), hematological adverse event (SAE), CMV infection, BK virus infection, MACE(major cardiac adverse event) and cancer

SECONDARY OUTCOMES:
Recipient Efficacy (any adverse events) | During one year
  comparison during the first year between the two groups for: patient and graft survival, delayed graft function, one year rate of acute rejection, occurrence od de novo DSA, renal function at one year (eGFR,MDRD)
Recipient Safety (any adverse events) | During one year
  Comparison during the first year between the two groups for various infections (virus, bacteria, fungi), hematological adverse event (SAE or not)
Reconstitution of the T, and B cell populations | During one year
  Reconstitution of the T, and B cell populations at D0, D7, M3, M12
Cost comparison | During one year
  Hospitals costs at 1 year months (including re-hospitalisation costs)

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Amiens Picardie, Hopital Sud, Amiens
  - CHU d'Angers, Angers
  - CHRU de Brest, Brest
  - CHU Hopital Clemenceau, Caen
  - CHU Hopital Gabriel Montpied, Clermont-Ferrand
  - CHU Dupuytren 2, Limoges
  - Hopital Necker Enfant Malade, Paris
  - CHU La Milétrie, Poitiers
  - CHU Hopital Maison Blanche, Reims
  - CHU de Rennes, Rennes
  - CHU Hopital de Bois Guillaume, Rouen
  - Hopitaux Universitaires de Strasbourg - Hopital civil, Strasbourg
  - CHRU de Tours, Tours